CLINICAL TRIAL: NCT02997969
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of HIV Clade C DNA and of MF59-adjuvanted Clade C Env Protein, in Healthy, HIV-uninfected Adult Participants
Brief Title: Safety and Immune Response to a Clade C DNA HIV Vaccine
Acronym: HVTN111
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); IPPOX Foundation (Other); Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 111
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: DNA + Placebo + Protein/MF59 (Active Comparator): Participants will receive the DNA-HIV-PT123 vaccine in the left deltoid at months 0, 1, 3, and 6. They will receive placebo in the right deltoid at months 0 and 1, and the Protein/MF59 vaccine at months 3 and 6. All injections are via needle and syringe.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Protein/MF59 vaccine; Biological: Placebo
- Group 2: DNA + Placebo + Protein/MF59 (Active Comparator): Participants will receive the DNA-HIV-PT123 vaccine in the left deltoid at months 0, 1, and 6. They will receive placebo in both deltoids at month 3, and the Protein/MF59 vaccine at months 0, 1, and 6. All injections are via needle and syringe.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Protein/MF59 vaccine; Biological: Placebo
- Group 3: Placebo (Placebo Comparator): Participants will receive placebo in both deltoids at months 0, 1, 3, and 6. All injections are via needle and syringe.
  Interventions: Biological: Placebo
- Group 4: DNA + Placebo + Protein/MF59 (Active Comparator): Participants will receive the DNA-HIV-PT123 vaccine via Biojector in the left deltoid at months 0, 1, 3, and 6. They will receive placebo in the right deltoid at months 0 and 1, and the Protein/MF59 vaccine at months 3 and 6, via needle and syringe.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Protein/MF59 vaccine; Biological: Placebo
- Group 5: DNA + Placebo + Protein/MF59 (Active Comparator): Participants will receive the DNA-HIV-PT123 vaccine at months 0, 1, and 6, and placebo at month 3, in the left deltoid via Biojector. They will receive placebo at month 3, and the Protein/MF59 vaccine at months 0, 1, and 6, in the right deltoid via needle and syringe.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Protein/MF59 vaccine; Biological: Placebo
- Group 6: Placebo (Placebo Comparator): Participants will receive placebo in the left deltoid via Biojector, and in the right deltoid via needle and syringe, at months 0, 1, 3, and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DNA-HIV-PT123 vaccine — Contains a mixture of 3 DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C ZM96 gag, 2) clade C ZM96 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose 4 mg administered as 1 mL intramuscularly (IM)
  Arms: Group 1: DNA + Placebo + Protein/MF59; Group 2: DNA + Placebo + Protein/MF59; Group 4: DNA + Placebo + Protein/MF59; Group 5: DNA + Placebo + Protein/MF59
Biological: Protein/MF59 vaccine — clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant, administered as 0.5 mL IM
  Other Names: Bivalent Subtype C gp120/MF59
  Arms: Group 1: DNA + Placebo + Protein/MF59; Group 2: DNA + Placebo + Protein/MF59; Group 4: DNA + Placebo + Protein/MF59; Group 5: DNA + Placebo + Protein/MF59
Biological: Placebo — Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products
  Other Names: Sodium Chloride, 0.9%

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to an HIV clade C DNA vaccine and to an MF59-adjuvanted clade C Env protein in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immunogenicity to DNA-HIV-PT123 (an HIV clade C DNA vaccine) and to Bivalent Subtype C gp120/MF59 in healthy, HIV-uninfected adults.

The study will enroll healthy, HIV-uninfected participants aged 18 to 40 years. Participants will be randomly assigned to one of 6 groups. Each group will receive experimental vaccine and protein and/or placebo at 4 study visits. Participants in Groups 1-3 will receive all injections via needle and syringe. Participants in Groups 4-6 will receive the DNA vaccine via Biojector, and protein and/or placebo via needle and syringe.

Participants in Groups 1 and 4 will receive the DNA vaccine at months 0, 1, 3, and 6 and the protein at months 3 and 6. Participants in Groups 2 and 5 will receive the DNA vaccine and the protein at months 0, 1, and 6 and placebo at month 3. Participants in Groups 3 and 6 will receive placebo at months 0, 1, 3, and 6.

Study visits will include a physical examination, an interview and/or questionnaire, HIV testing and HIV risk-reduction counseling, and urine and blood collection. Participants may optionally choose to provide rectal fluid, cervical fluid, or semen samples.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 40 years
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; provides answers to a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values:

Hemogram/Complete blood count (CBC)

* Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
* White blood cell count = 3,300 to 12,000 cells/mm^3
* Total lymphocyte count ≥ 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets = 125,000 to 550,000/mm^3 Chemistry
* Chemistry panel: ALT, AST, and ALP < 1.25 times the institutional upper limit of normal; creatinine ≤ institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive Urine
* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.

Reproductive status: A volunteer who was born female must:

* Agree to consistently use effective contraception (Appendix B) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit.

  * Effective contraception is defined as using 1 of the following methods:
  * Condoms (male or female), or
  * Diaphragm or cervical cap,
  * PLUS 1 of the following methods:
  * Intrauterine device (IUD),
  * Hormonal contraception (in accordance with applicable national contraception guidelines),
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity after vasectomy); or
  * Any other contraceptive method approved by the HVTN 111 PSRT
* Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
* Or be sexually abstinent. Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit Other Volunteers 21 years of age and older who were born female consenting to provide cervical samples: pap smear within the 3 years prior to enrollment, with the latest result reported as normal or ASCUS (atypical squamous cells of undetermined significance); for those 21 years and older that have not had a pap smear within the last 3 years prior to enrollment, must be willing to undergo a pap smear with the result reported as normal or ASCUS prior to sample collection.

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 111 study
* Pregnant or breastfeeding Vaccines and other Injections
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 111 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 111 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 111 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination Immune System
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded from participation: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines or to vaccine components such as eggs, egg products, or neomycin, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency Clinically significant medical conditions
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Frequency of severe local and systemic reactogenicity signs and symptoms (pain, tenderness, erythema, induration, fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia) | Measured through Month 12
Frequency of adverse events (AEs) | Measured through Month 12
  By body system, Medical Dictionary for Regulatory Activities (MedDRA) preferred term, severity, and assessed relationship to study products
Frequency of serious adverse events (SAEs), adverse events of special interest (AESIs), and new chronic conditions (requiring medical intervention for 30 days or more) | Measured through Month 12
Composite of safety laboratory measures: white blood cells (WBC), neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphate (ALP), and creatinine | Measured through Month 12
Frequency of AEs leading to early participant withdrawal or early discontinuation of study products administration | Measured through Month 12
HIV-specific total immunoglobulin G (IgG) binding antibody response breadth and magnitude as assessed by multiplex assay | Measured through Month 6.5
Anti-V1/V2 scaffold IgG binding antibody responses as assessed by multiplex assay | Measured through Month 6.5
Presence of neutralizing antibody responses against HIV-1 isolates | Measured through Month 6.5
HIV-specific CD4+ T-cell responses as assessed by flow cytometry | Measured through Month 6.5
HIV-specific CD8+ T-cell responses as assessed by flow cytometry | Measured through Month 6.5

CONTACTS AND LOCATIONS:
Overall Officials: Mina Hosseinipour, Study Chair — UNC Project- Lilongwe
Locations (5):
- South Africa (3):
  - Aurum Tembisa CRS, Johannesburg, Gauteng
  - Isipingo CRS, Westville, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) Network CRS, Mbeya, Tanzania
- Matero Reference Clinic CRS, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Hanass-Hancock J, Carpenter B, Reddy T, Nzuza A, Gaffoor Z, Goga A, Andrasik M. Participants' characteristics and motivations to screen for HIV vaccine and monoclonal antibody trials in KwaZulu-Natal, South Africa. Trials. 2021 Dec 11;22(1):897. doi: 10.1186/s13063-021-05792-7. PMID 34895272
- [Derived] Hosseinipour MC, Innes C, Naidoo S, Mann P, Hutter J, Ramjee G, Sebe M, Maganga L, Herce ME, deCamp AC, Marshall K, Dintwe O, Andersen-Nissen E, Tomaras GD, Mkhize N, Morris L, Jensen R, Miner MD, Pantaleo G, Ding S, Van Der Meeren O, Barnett SW, McElrath MJ, Corey L, Kublin JG; HVTN 111 Protocol Team. Phase 1 Human Immunodeficiency Virus (HIV) Vaccine Trial to Evaluate the Safety and Immunogenicity of HIV Subtype C DNA and MF59-Adjuvanted Subtype C Envelope Protein. Clin Infect Dis. 2021 Jan 23;72(1):50-60. doi: 10.1093/cid/ciz1239. PMID 31900486